CLINICAL TRIAL: NCT01516632
Title: Smoking Cessation Via Text Messaging: Feasibility Testing of SMS USA
Brief Title: Smoking Cessation Via Text Messaging: Feasibility Testing of Stop My Smoking USA
Acronym: SMS USA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: Michigan State University (Other); The University of Texas Health Science Center, Houston (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21CA135669 (NIH); 5R21CA135669 (NIH)
Record Dates: First submitted 2011-03-15; First posted 2012-01-25 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: Smoking Cessation
Keywords: Cellular Phone; Mobile Phone; Cognitive Behavior Therapy; Technology; Smoking cessation; young adults
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS USA (Experimental): The 6-week smoking cessation intervention
  Interventions: Behavioral: SMS USA
- Attention matched control (No Intervention): Messages aimed at improving one's sleep and increasing one's fitness, along with general messages about the most well known health dangers of smoking. Messages sent on the same schedule as the intervention group.

INTERVENTIONS:
Behavioral: SMS USA — Intervention participants receive text messages daily pre-and post-quit. Everyone receives messages 14 days prior to the Quit day, and through the day after Quit. Then, participants are 'pathed' to particular messages based upon their self-reported smoking status at Day 2 and Day 7 post quit, respectively. Those who are successful at quitting receive messages aimed at relapse prevention whereas those who have slipped receive messages aimed at getting the person to recommit to quitting and trying again.
  Other Names: Stop My Smoking USA
  Arms: SMS USA

SUMMARY:
The investigators developed a text messaging-based smoking cessation program called SMS (Stop My Smoking) USA. It was tailored for the unique needs and smoking habits of young adults. The investigators hypothesized that those in the SMS USA intervention would be significantly more likely to be quit at 6-months compared to the attention-matched control group.

DETAILED DESCRIPTION:
About one in four young adults are current smokers. Although over half report the desire to quit or cut down, quit rates in this age group have remained stagnant in the last ten years. Text messaging may represent a compelling intervention delivery method for smoking cessation for young adults because it is a medium they have widely adopted. Cell phone interventions also are unique because of their 'always on' capability - interventions are never far from the young adult's reach and they are received automatically instead of requiring the participant to initiate contact in order to receive the information. Dr. Ybarra, along with Drs. Holtrop and Graham, have developed SMS Turkey, an innovative behavioral intervention that uses text messaging to deliver CBT-based smoking cessation information to participants daily. Successful use of text messaging to deliver smoking cessation programs has been reported by Rodgers and colleagues in New Zealand and a replication study they are leading in the United Kingdom. These data provide optimism for the feasibility of text messaging-based smoking cessation programs in the United States. Using qualitative methods to inform design and content, and quantitative methods to assess the feasibility of the program, we propose to design and test SMS (Stop My Smoking) USA, a cell-phone based smoking cessation program for young adults ages 18-25. This innovative smoking cessation program uses technology widely adopted by young adults, an under-targeted population, to deliver a proactive, cognitive behavioral therapy (CBT)-based intervention. Our multidisciplinary team of researchers brings together expertise in Internet health and the design of tailored smoking cessation interventions.

ELIGIBILITY:
Inclusion Criteria:

* 28 cigarettes or more per week (at least 4/day) and on at least 6 days/week.
* Owning a text-capable cell phone and cognizant of how to send and receive text messages
* Currently enrolled or intending to enroll in an unlimited text messaging plan
* Enrolled with a cell phone carrier that was compatible with the program software
* Agree to verification of smoking cessation status by a significant other
* Able to read and write in English
* Informed consent

Exclusion Criteria:

None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ybarra, MPH PhD, Principal Investigator — Center for Innovative Public Health Research
Locations (1):
- Internet Solutions for Kids, Inc., Santa Ana, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ybarra ML, Holtrop JS, Prescott TL, Strong D. Process evaluation of a mHealth program: lessons learned from Stop My Smoking USA, a text messaging-based smoking cessation program for young adults. Patient Educ Couns. 2014 Nov;97(2):239-43. doi: 10.1016/j.pec.2014.07.009. Epub 2014 Jul 17. PMID 25103183
- [Background] Ybarra ML, Prescott TL, Holtrop JS. Steps in tailoring a text messaging-based smoking cessation program for young adults. J Health Commun. 2014 Dec;19(12):1393-407. doi: 10.1080/10810730.2014.901441. Epub 2014 Apr 25. PMID 24766267
- [Background] Filion AJ, Darlington G, Chaput JP, Ybarra M, Haines J. Examining the influence of a text message-based sleep and physical activity intervention among young adult smokers in the United States. BMC Public Health. 2015 Jul 16;15:671. doi: 10.1186/s12889-015-2045-2. PMID 26178640
- [Result] Ybarra ML, Holtrop JS, Prescott TL, Rahbar MH, Strong D. Pilot RCT results of stop my smoking USA: a text messaging-based smoking cessation program for young adults. Nicotine Tob Res. 2013 Aug;15(8):1388-99. doi: 10.1093/ntr/nts339. Epub 2013 Jan 24. PMID 23348969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited nationally through online advertisements (e.g. Craigslist) between May 3, 2011 and August 4, 2011. Smokers expressed their interest by completing an online screener form, which was then e-mailed to the project coordinator.
Pre-assignment Details: Of the 1,916 people who expressed interest, 585 (31%) were eligible for the study. Of these 585, contact was not made with 49% (n = 284). Fifteen percent (n=90) declined to participate. 211 eligible participants consented to participate and were randomized into the study. 47 terminated after randomization (i.e. did not complete enrollment process)
Groups:
- Smoking Cessation Text Messaging: 6-week smoking cessation program delivered via daily text messages. Stop My Smoking (SMS) USA is a text messaging-based smoking cessation program tailored to the experiences of young adult smokers. Content was tailored based on participant's stage of quitting (i.e. pre-quit, quit day, early-quit, late-quit, relapse). Based on the typical trajectory, content paths were created for participants based on whether or not they were smoking 2 days after quit day; and again at 7 days after quit day. The intervention group had access to Text Buddy (another person in the program that a participant was assigned to so they could text one another for support anonymously and Text Crave (immediate, on demand messages aimed at helping the participant through a craving).
- Attention-Matched Control Group: Control group participants received a text-messaging program that was similar to the intervention program on the number of text messages received per day across the 6 weeks. Message content was aimed at improving one's sleep and exercise habits within the context of how it would help the participant quit smoking. Messages were not tailored based on quitting stage (e.g., Pre-Quit vs. Early Quit) nor were Text Buddy and Text Crave components available to this group.
Period: Overall Study
Arm/Group | Smoking Cessation Text Messaging | Attention-Matched Control Group
Started | 101 | 63
Completed | 77 | 48
Not Completed | 24 | 15

BASELINE CHARACTERISTICS:
Groups:
- The Control Group: Control group participants received a text-messaging program that was similar to the intervention program on the number of text messages received per day across the 6 weeks. Message content was aimed at improving one's sleep and exercise habits within the context of how it would help the participant quit smoking. Messages were not tailored based on quitting stage (e.g., Pre-Quit vs. Early Quit) nor were Text Buddy and Text Crave components available to this group.
- Total: Total of all reporting groups
Arm/Group | Smoking Cessation Text Messaging | The Control Group | Total
Number analyzed (Participants) | 101 | 63 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.6 (2.1) | 21.6 (2.1) | 21.6 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 28 | 72
  Male | 57 | 35 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 8 | 30
  Not Hispanic or Latino | 79 | 55 | 134
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 13 | 9 | 22
  White | 65 | 41 | 106
  More than one race | 16 | 8 | 24
  Unknown or Not Reported | 4 | 0 | 4
Average number of cigarettes smoke per day [Mean (Standard Deviation); unit: number of cigarettes per day] | 12.4 (6.3) | 11.9 (5.7) | 12.2 (6.1)
Nicotine dependent [Number; unit: participants]
  Yes | 90 | 59 | 149
  No | 11 | 4 | 15
Importance of Quitting [Mean (Standard Deviation); unit: units on a scale] — The score ranged from 0-10 with higher scores reflecting more importance Miller, W. R., Zweben, A., DiClemente, C. C., & Rychtarik, R. G. (1992). Motivational Enhancement Therapy Manual: A clinical research guide for therapists treating individuals with alcohol abuse and dependence. Rockville, MD: National Institute on Alcohol Abuse and Alcoholism.
  units on a scale | 8.7 (1.5) | 8.9 (1.3) | 8.8 (1.4)
Confidence of one's ability to quit [Mean (Standard Deviation); unit: units on a scale] — The score ranged from 0-10 with higher scores reflecting more confidence Miller, W. R., Zweben, A., DiClemente, C. C., & Rychtarik, R. G. (1992). Motivational Enhancement Therapy Manual: A clinical research guide for therapists treating individuals with alcohol abuse and dependence. Rockville, MD: National Institute on Alcohol Abuse and Alcoholism.
  units on a scale | 6.7 (2.2) | 6.5 (2.6) | 6.6 (2.4)
Income [Number; unit: participants] — Low Income is <$35,000
  participants
    <$35,000 | 85 | 57 | 142
    >$35,000 | 16 | 6 | 22
Married/living with someone [Number; unit: participants]
  Yes | 29 | 17 | 46
  No | 72 | 46 | 118
Current Employment Status [Number; unit: participants]
  Not Working | 36 | 35 | 71
  Working ≤ 30 hr | 24 | 12 | 36
  Working > 30 hr | 41 | 16 | 57
Currently Enrolled in College, University, or Junior College [Number; unit: participants]
  Yes | 43 | 25 | 68
  No | 58 | 38 | 96
Tenure with current cell phone number (months) [Mean (Standard Deviation); unit: Months] — The length of time they have had the current cellular phone number
  Months | 44.8 (28.2) | 46.4 (31.6) | 45.4 (29.5)
Number of text messages sent on an average day [Median (Inter-Quartile Range); unit: units on a scale] | 50 [20 to 100] | 45 [20 to 100] | 50 [20 to 100]
Number of text messages received on an average day [Median (Inter-Quartile Range); unit: text messages per day] | 60 [20 to 100] | 50 [18 to 100] | 50 [20 to 100]
Planning on using an evidence-based quitting aid [Number; unit: participants] — Planning on using an evidence-based quitting aid for the current attempt
  participants
    Yes | 26 | 11 | 37
    No | 75 | 52 | 127
Resistance self-efficacy [Mean (Standard Deviation); unit: units on a scale] — The scale was a 4-item measure developed by Lawrance L, Rubinson L. Self-efficacy as a predictor of smoking behavior in young adolescents. Addict Behav. 1986;11(4):367-382.
  The possible range of scores was from 4-20 with higher scores reflecting more self-efficacy.
  units on a scale | 10.6 (4.0) | 10.5 (4.0) | 10.55 (4.0)
Social support from "special person" [Mean (Standard Deviation); unit: units on a scale] — Measured using the Multidimensional Scale of Perceived Social Support (Zimet, Dahlem, Zimet, & Farley, 1988)
  The values range 4-20 with higher scores reflecting more social support
  units on a scale | 15.1 (5.4) | 16.3 (3.9) | 15.6 (4.9)
Social support from friends [Mean (Standard Deviation); unit: units on a scale] — Measured using the Multidimensional Scale of Perceived Social Support (Zimet, Dahlem, Zimet, & Farley, 1988)
  The values range 4-20 with higher scores reflecting more social support
  units on a scale | 16.1 (4.0) | 16.6 (3.1) | 16.3 (3.7)
Social support from family [Mean (Standard Deviation); unit: units on a scale] — Measured using the Multidimensional Scale of Perceived Social Support (Zimet, Dahlem, Zimet, & Farley, 1988)
  The values range 4-20 with higher scores reflecting more social support
  units on a scale | 15.3 (4.3) | 15.9 (3.6) | 15.5 (4.1)
Depressive Symptomatology [Mean (Standard Deviation); unit: units on a scale] — Center for Epidemiologic Studies Depression Scale (Eaton, Muntaner, Smith, Tien, & Ybarra, 2004)
  The scores range 0-27 with higher scores reflecting more depressive symptomatology
  units on a scale | 7.8 (6.2) | 9.3 (6.4) | 8.3 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Continuous Abstinence at 3-months Assessed in Accordance With the NIH Behavior Change Consortium's Recommendations
Description: Continuous abstinence is defined as 5 or fewer cigarettes smoked since one's quit date. The question was asked based upon West et al., 2005: "Have you smoked at all, even just a puff, since [insert quit date]?" If yes, the respondent will be probed for how many cigarettes were smoked. Responses will be categorized into one of three options: A) No, not a puff; B) 1-5 cigarettes; C) More than 5 cigarettes.
  Self-reported cessation is confirmed by a significant other.
Time Frame: 3-months post-quit
Measure: Number; unit: participants
Groups:
- Smoking Cesssation Via Text Messaging: The 6-week smoking cessation program
  SMS (Stop my Smoking) USA: Intervention participants receive text messages daily pre-and post-quit. Everyone receives messages 14 days prior to the Quit day, and through the day after Quit. Then, participants are 'pathed' to particular messages based upon their self-reported smoking status at Day 2 and Day 7 post quit, respectively. Those who are successful at quitting receive messages aimed at relapse prevention whereas those who have slipped receive messages aimed at getting the person to recommit to quitting and trying again.
- Attention Matched Control: Messages aimed at improving one's sleep and increasing one's fitness, along with general messages about the most well known health dangers of smoking. Messages sent on the same schedule as the intervention group.
  SMS (Stop my Smoking) USA: Intervention participants receive text messages daily pre-and post-quit. Everyone receives messages 14 days prior to the Quit day, and through the day after Quit. Then, participants are 'pathed' to particular messages based upon their self-reported smoking status at Day 2 and Day 7 post quit, respectively. Those who are successful at quitting receive messages aimed at relapse prevention whereas those who have slipped receive messages aimed at getting the person to recommit to quitting and trying again.
Arm/Group | Smoking Cesssation Via Text Messaging | Attention Matched Control
Number analyzed (Participants) | 101 | 63
participants | 40 | 19
Statistical Analysis 1: Comparison: Smoking Cesssation Via Text Messaging vs Attention Matched Control; Test type: Superiority or Other; Odds Ratio (OR) = 1.62, 95% CI 2-sided [.82 to 3.21]

2. Secondary Outcome: Point Prevalence
Description: A cigarette, even just a puff, within the last 7 days (yes/no).
Time Frame: 4-weeks post-quit
Measure: Number; unit: participants
Arm/Group | Smoking Cessation Text Messaging | Attention-Matched Control Group
Number analyzed (Participants) | 101 | 63
participants | 44 | 17
Statistical Analysis 1: Comparison: Smoking Cessation Text Messaging vs Attention-Matched Control Group; Test type: Superiority or Other; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.22 to 5.30]

3. Secondary Outcome: Continuous Abstinence at 4-weeks Post-quit
Description: Smoking five or fewer cigarettes since quit day at 4 weeks post-quit as verified by a significant other
Time Frame: 4 weeks post-quit
Measure: Number; unit: participants
Arm/Group | Smoking Cessation Text Messaging | Attention-Matched Control Group
Number analyzed (Participants) | 101 | 63
participants | 34 | 13
Statistical Analysis 1: Comparison: Smoking Cessation Text Messaging vs Attention-Matched Control Group; Test type: Superiority or Other; Odds Ratio (OR) = 3.33, 95% CI 2-sided [1.48 to 7.45]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the study period (i.e., from baseline to 4-week follow-up)
Arm/Group | Smoking Cessation Text Messaging | Attention-Matched Control Group
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/63
Other Adverse Events (participants affected / at risk) | 0/101 | 0/63

LIMITATIONS AND CAVEATS:
The main limitation of the study is its small sample size. Also, it is unclear how young adult smokers recruited on Craigslist compared with young adult smokers who would be recruited through other ways.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No